CLINICAL TRIAL: NCT02319655
Title: Changes of the Subfoveal Hyporeflective Zone After Membrane Peeling With Air Tamponade and Balanced Salt Solution - a Pilot Study
Brief Title: Morphologic Changes After Membrane Peeling With Air Tamponade and Balanced Salt Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim.Prof.Dr.MBA, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP; EK-14-013-0214 (Other: Ethikkommission der Stadt Wien)
Record Dates: First submitted 2014-06-02; First posted 2014-12-18 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Epiretinal Membrane; Macular Pucker
Keywords: Epiretinal membrane; Macular pucker; Membrane peeling; pars plana vitrectomy; Air; balanced salt solution; Intraoperative OCT; Hyporeflectivity; Retina
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air tamponade (Active Comparator): Air is injected after vitrectomy/membrane peeling
  Interventions: Procedure: Air tamponade
- Balanced salt solution filling (Active Comparator): Balances salt solution is injected after vitrectomy/membrane peeling
  Interventions: Procedure: Balanced salt solution filling

INTERVENTIONS:
Procedure: Air tamponade — Air tamponade
  Arms: Air tamponade
Procedure: Balanced salt solution filling — BSS filling
  Arms: Balanced salt solution filling

SUMMARY:
During the last decade optical coherence tomography (OCT) extended the possibilities for in vivo macula diagnostic and was increasingly used for pre- and post-operative imaging of retinal diseases. Spectral-domain optical coherence tomography (SD-OCT) with its increased scanning speed and image-resolution provides more detailed information of microstructures in the macula. Epiretinal membrane (ERM) is a disorder involving the posterior pole of the eyeball. It can be idiopathic or caused secondarily in various ocular conditions, such as uveitis, trauma, retinal detachment or retinal vascular diseases. In patients who suffer from loss of vision and metamorphopsia, vitrectomy and membrane peeling is usually performed to remove the ERM.

Different study groups showed that intraoperative use of SD-OCT is possible. Two groups already achieved to work operation microscope integrated SD-OCT setup. Due to the high axial resolution of the SD-OCT some groups reported about an increased hyporeflective zone in the subfoveal region appearing directly after the membrane peeling procedure. It was hypothesized that this phenomenon could be an expression of surgical trauma, as this hyporeflective zone disappears in follow up OCT 10 days after surgery.

DETAILED DESCRIPTION:
During the last decade optical coherence tomography (OCT) extended the possibilities for in vivo macula diagnostic and was increasingly used for pre- and post-operative imaging of retinal diseases. Spectral-domain optical coherence tomography (SD-OCT) with its increased scanning speed and image-resolution provides more detailed information of microstructures in the macula. Epiretinal membrane (ERM) is a disorder involving the posterior pole of the eyeball. It can be idiopathic or caused secondarily in various ocular conditions, such as uveitis, trauma, retinal detachment or retinal vascular diseases. In patients who suffer from loss of vision and metamorphopsia, vitrectomy and membrane peeling is usually performed to remove the ERM.

Different study groups showed that intraoperative use of SD-OCT is possible. Two groups already achieved to work operation microscope integrated SD-OCT setup. Due to the high axial resolution of the SD-OCT some groups reported about an increased hyporeflective zone in the subfoveal region appearing directly after the membrane peeling procedure. It was hypothesized that this phenomenon could be an expression of surgical trauma, as this hyporeflective zone disappears in follow up OCT 10 days after surgery .

The aim of the study is to use a microscope integrated SD-OCT in order to measure the surgically induced hyporeflective zone in the subfoveal region during membrane peeling and to evaluate whether the hyporeflective zone, that is believed to be an expression of tissue trauma, disappears faster with air tamponade compared to eyes with balanced saline solution (BSS).

Both, intraocular air tamponade and BSS are commonly used after vitrectomy with membrane peeling and pose the standard of care for this operation and no information concerning the superiority of one method is available. The non-contact microscope integrated SD-OCT, does not require any relevant additional time during the operation procedure (max. 2 minutes per operation for the OCT scans). During the OCT measurement time the light of the microscope will be reduced to a minimum to avoid additional light exposure. The OCT scans will be performed only at different time points (as mentioned below) to keep the OCT light exposure low and far below the acceptable exposure time as mentioned in the OCT safety guidelines.

SD-OCT is a safe and commonly used diagnostic tool in ophthalmology and its application does not bear any additional risk for the patients included in the study. Furthermore, all devices used in this study are CE-marked (Communauté Européenne).

Patients included in this study will not have a direct benefit from participation. However, it is very likely that the evaluation of the hyporeflective zone is the main indicator for the postoperative visual quality of a patient and this study will help to clarify, if air, or BSS have a protective effect for the fovea. In consequence, this study should help to use an intra-operative treatment that leads to a faster visual rehabilitation after membrane peeling.

ELIGIBILITY:
Inclusion Criteria:

* Epiretinal membrane and the indication for surgery (visual symptoms)
* Age 21 and older
* written informed consent prior to surgery

Exclusion Criteria:

* Patients who have already undergone vitrectomy
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Proportion of eyes with presence of a hyporeflective zone on the 7th postoperative day on OCT scan | 7 days postoperatively
  An expert in the field of reading retinal OCT scans will assess whether or not a hyporeflective zone on the 7th postoperative day is visible on the OCT scan

SECONDARY OUTCOMES:
Change in retinal thickness 3 months after surgery assessed with OCT | 3 months
  Central retinal thickness assessed with OCT (µm)
Attachment of the posterior hyaloid membrane before starting surgery assessed with intraoperative OCT | intraoperatively
  An expert in the field of reading retinal OCT scans will assess intraoperative OCT scans and determine whether or not the posterior hyaloid membrane is attached to the retina before initiation of the surgery.
Best corrected visual acuity | 3 months postoperatively
  ETDRS (Early treatment of diabetic retinopathy study) reading charts will be used to assess best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD,Prof,MBA, Principal Investigator — VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital Vienna, Vienna, Austria 1140
Locations (1):
- Oliver Findl, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided